CLINICAL TRIAL: NCT04809428
Title: The Use of vNOTES Approach in Elective Bilateral Salpingectomy for Sterilization as a Cancer Prevention Strategy
Brief Title: vNOTES in Elective Bilateral Salpingectomy for Sterilization
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, Principal investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: vNOTES Salpingectomy
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Sterility, Female
Keywords: vNOTES; Scarless surgery; cancer prevention
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vNOTES Salpingectomy: Elective bilateral salpingectomy by vaginal Natural Orifice Transluminal Endoscopic Surgery approach
  Interventions: Procedure: vNOTES salpingectomy
- LS Salpingectomy: Elective bilateral salpingectomy by conventional laparoscopy
  Interventions: Procedure: Laparoscopic salpingectomy

INTERVENTIONS:
Procedure: vNOTES salpingectomy — Surgical removal of both salpinx by vNOTES with using a 3-cm of posterior colpotomy and either glove port or Gel point V path. Colpotomy will be closed with using 2.0 rapid vicryl.
  Groups: vNOTES Salpingectomy
Procedure: Laparoscopic salpingectomy — Surgical removal of both salpinx by conventional laparoscopy in a standardised fashion: with using one 10-mm umbilical and two 5-mm lateral ports.
  Groups: LS Salpingectomy

SUMMARY:
Objective: To compare the vNOTES approach versus conventional laparoscopic approach to be used in elective bilateral salpingectomy for sterilisation as an opportunistic cancer prevention strategy.

Study design: Prospective cohort, two-centred trial. Study population: All women aged over 18 who are planned to undergo for definitive surgical sterilisation regardless of parity with a non-prolapsed uterus.

Primary outcomes: (1) Patient satisfaction (at 1st week and 1st month of the surgery) measured by The Patient Global Imression of Improvement (PGI-I), (2) Postoperative early pain (Visual Analog Score (VAS) at 6th and 24th hours of the surgery).

Secondary outcomes: (1) Conversion to laparoscopy or laparotomy, (2) duration of the procedure, (3)total amount of analgesics used, (4) New-onset dyspareunia at first coitus measured by the Pain subdomain of Female Sexual Function Index (FSFI), (5) intraoperative complications, (6) postoperative complications

DETAILED DESCRIPTION:
Women who are indicated or seek for surgical sterilisation are routinely offered salpingectomy rather than tubal ligation for cancer prevention purposes as a local protocol. Those patients will be offered for vNOTES approach after detailed patient counselling and will be enrolled to the study upon acceptation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18 years regardless of parity with a non-prolapsed uterus
* Patients who are indicated or seek for definitive surgical sterilisation
* Patients who prefers salpingectomy over tubal ligation after considering its possible cancer prevention effect
* Written informed consent obtained prior to surgery

Exclusion Criteria:

* Any malignancy
* Suspected rectovaginal endometriosis
* History of pelvic inflammatory disease, pouch of Douglas abscess
* Being Virgo or Pregnant
* Failure to provide written informed consent prior to surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women seeking for definitive surgical sterilization who prefers salpingectomy over tubal ligation due to its possible cancer risk reduction effect.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction at first week | The first week after the surgical procedure
  Patient satisfaction will be measured with Patient Global Impression of Improvement (PGI-I). It is scored as: Very much better (1), Much better (2), A little better (3), No change (4), A little worse (5), Much worse (6), Very much worse (7). Patient reported as Very much better or much better will be regarded as satisfied.
Patient satisfaction at first month | The first month after the surgical procedure
  Patient satisfaction will be measured with Patient Global Impression of Improvement (PGI-I). It is scored as: Very much better (1), Much better (2), A little better (3), No change (4), A little worse (5), Much worse (6), Very much worse (7). Patient reported as Very much better or much better will be regarded as satisfied.
Postoperative pain at 6th hours | At the 6th hours after the surgical procedure
  Postoperative pain scores will be measured with using Visual Analogue Score (VAS) as self-reported by the participating women. The VAS scores range from 0= no pain to 10= worst imaginable pain.
Postoperative pain at 24th hours | At the 24th hours after the surgical procedure
  Postoperative pain scores will be measured with using Visual Analogue Score (VAS) as self-reported by the participating women. The VAS scores range from 0= no pain to 10= worst imaginable pain.

SECONDARY OUTCOMES:
Dyspareunia | At 1st month after the surgical procedure
  Subjective Success - Change from baseline Female Sexual Function Index (FSFI) to measure sexual dysfunction at first month.
  Validated into Turkish language form will be used to compare preoperative and postoperative period. The FSFI is a multiple-trait scoring, self-report document used to assess female sexual function. It consists of 19 items that encompass six separate domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The maximum score is 36 points and the minimum score is 2 points. Only pain subdomain will be used for research purposes.
Duration of the surgical procedure | Intraoperative
  Duration of the surgery will be measured in minutes, in between the first vaginal/abdominal incision and vaginal/abdominal wound closure.
Conversion | Intraoperative
  Conversion to laparoscopy or laparotomy will be noted.
Need of Analgesics | Postoperative, 24 hours
  Patients will not be routinely offered additional analgesics and the need of additional analgesics will be noted if patient desires for.
Intraoperative complications | Intraoperative
  Any minor and major (e.g., bowel injury, bleeding>300cc, major vessel injury) complications that occur during the surgery
Postoperative complications | Postoperative, in the first month of the surgery
  Any minor and major complications (e.g., bowel injury, haematoma, infection, dyspareunia, vaginal pain, sexual discomfort) that occur in the first month of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Kaya, MD, Principal Investigator — Bakirkoy Sadi Konuk Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Bakirkoy Sadi Konuk Training and Research Hospital, Istanbul
  - Sehit Prof Dr Ilhan Varank Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Upon request, after the work is published
Supporting Information: CSR
Time Frame: Upon request, after the work is published, 5 years
Access Criteria: Upon request, after the work is published, 5 years

REFERENCES:
- [Background] Kaya C, Alay I, Cengiz H, Baghaki S, Aslan O, Ekin M, Yasar L. Conventional Laparoscopy or Vaginally Assisted Natural Orifice Transluminal Endoscopic Surgery for Adnexal Pathologies: A Paired Sample Cross-Sectional Study. J Invest Surg. 2021 Nov;34(11):1185-1190. doi: 10.1080/08941939.2020.1789246. Epub 2020 Jul 7. PMID 32633168
- [Background] Yassa M, Pulatoglu C. Patients' perceptions toward and the driving factors of decision-making for opportunistic bilateral salpingectomy at the time of cesarean section. Turk J Obstet Gynecol. 2020 Jun;17(2):115-122. doi: 10.4274/tjod.galenos.2020.12129. Epub 2020 Jul 29. PMID 32850186
- [Background] Kaya C, Alay I, Yildiz S, Cengiz H, Afandi X, Yasar L. The Feasibility of Natural Orifice Transluminal Endoscopic Surgery in Gynecology Practice: Single-Surgeon Experience. Gynecol Minim Invasive Ther. 2020 Apr 28;9(2):69-73. doi: 10.4103/GMIT.GMIT_84_19. eCollection 2020 Apr-Jun. PMID 32676283
- [Background] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BWJ, Bosteels JJA. Transvaginal natural orifice transluminal endoscopic surgery (vNOTES) adnexectomy for benign pathology compared with laparoscopic excision (NOTABLE): a protocol for a randomised controlled trial. BMJ Open. 2018 Jan 10;8(1):e018059. doi: 10.1136/bmjopen-2017-018059. PMID 29326183
- [Derived] Yassa M, Kaya C, Kalafat E, Tekin AB, Karakas S, Mutlu MA, Birol P, Tug N. The Comparison of Transvaginal Natural Orifice Transluminal Endoscopic Surgery and Conventional Laparoscopy in Opportunistic Bilateral Salpingectomy for Permanent Female Sterilization. J Minim Invasive Gynecol. 2022 Feb;29(2):257-264.e1. doi: 10.1016/j.jmig.2021.08.009. Epub 2021 Aug 16. PMID 34411729